CLINICAL TRIAL: NCT02133521
Title: Addition of DLBS1033 to Standard Therapy for Acute Ischemic Stroke Patients
Brief Title: DLBS1033 for Acute Ischemic Stroke Patients
Acronym: ADDLIST
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Very low recruitment rate. The Study Sites classified as tertiary referral hospital. Therefore, patients being referred to the site are mostly those with comorbidities included in the exclusion criteria.
Sponsor: Dexa Medica Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DLBS1033-0111
Record Dates: First submitted 2014-05-07; First posted 2014-05-08 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Acute Ischemic Stroke; Partial Anterior Circulation Infarct; Lacunar Anterior Circulation Infarct
Keywords: DLBS1033; Acute ischemic stroke; NIHSS; Barthel Index
MeSH Terms: conditions — Ischemic Stroke | interventions — DLBS 1033

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo 3 x 1 tablet, given everyday for 28 days of study period
  Interventions: Drug: Placebo
- DLBS1033 (Experimental): DLBS1033 enteric-coated tablet 3 x 490 mg daily, given everyday for 28 days of study period
  Interventions: Drug: DLBS1033

INTERVENTIONS:
Drug: DLBS1033 — Investigational drug or placebo will be given in addition to the standard therapy, consists of: aspirin enteric-coated tablet 1 x 80 mg daily, simvastatin film-coated tablet 1 x 20 mg daily, and vitamin B complex 1 x 1 tablet
  Other Names: Disolf
  Arms: DLBS1033
Drug: Placebo — Investigational drug or placebo will be given in addition to the standard therapy, consists of: aspirin enteric-coated tablet 1 x 80 mg daily, simvastatin film-coated tablet 1 x 20 mg daily, and vitamin B complex 1 x 1 tablet
  Arms: Placebo

SUMMARY:
This is a prospective, randomized, double-blind, and controlled clinical study to investigate the effects of DLBS1033 in conjunction with standard therapy compared to standard therapy alone in acute ischemic stroke patients. It is hypothesized that the improvement in functional outcomes as measured by NIHSS and BI as well as the improvement in haemostatic parameters as measured by thrombocyte aggregation test (TAT), fibrinogen, and d-dimer in DLBS group will be significantly greater than those in the control group.

DETAILED DESCRIPTION:
Subjects in this study will be screened consecutively and eligible subjects will be randomized into two groups and receive the investigational drug, DLBS1033 at a dose of 490 mg three times daily or its placebo in addition to standard therapy for 28-days course of therapy. Standard therapy used in this study will consist of: aspirin 80 mg, simvastatin 20 mg, and vitamin B complex.

After hospital admission and diagnosis, patient will be handled as per acute ischemic stroke management in each study site. Right after the patient is confirmed eligible to the study, the treatment(s) will be switched immediately into the study treatments. Clinical and laboratory examinations to evaluate the investigational drug's efficacy will be performed at baseline and 3, 7,14, and 28 days after study medication initiation; while safety examinations will be performed at the same time point, but 3 and 14 days after study medication initiation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent from the patients or patients' legally acceptable representatives (must be obtained before any trial related activities).
* Male or female subjects with age of >18 years at Screening.
* Patients clinically diagnosed having acute ischemic stroke attack and confirmed by CT scan.
* Patients with cerebral infarction subtypes of PACI or LACI as classified by Bamford criteria.
* Patients with moderate condition based on National Institutes of Health Stroke Scale (NIHSS) score of 5-15.
* Patients present at hospital and receiving first dose of study medication within 72 hours after the onset of the stroke symptoms.
* Able to take oral medication.

Exclusion Criteria:

* For females of childbearing potential: pregnancy and lactation period.
* History of hemorrhagic stroke within the last 3 months.
* Patients with seizure at the onset of stroke or with regular medication for seizure/epilepsy.
* Current or regular use (within the last 1 month) of oral anticoagulants, antiplatelets other than study medication, and herbal medicines.
* Patients who have received tissue plasminogen activator (TPA) within 24 hours to Screening.
* History of serious head injury within the last 3 months.
* History of major surgery within the last 3 months.
* Recent serious cardiovascular conditions, such as myocardial infarction and heart atrial fibrillation as demonstrated by electrocardiography (ECG).
* History of congestive heart failure and aortic dissection.
* Presence of severe renal and hepatic dysfunction, defined as serum creatinine level > 3x upper limit of normal (ULN) or history of hemodialysis, and any of serum ALT, AST, Gamma-GT level of > 3x ULN, respectively.
* Presence of acute SIRS.
* Presence of chronic infections.
* Patients with higher risks of bleeding.
* Subjects with uncontrolled hypertension (systolic blood pressure > 185 mmHg or diastolic blood pressure > 110 mmHg).
* Subjects with random plasma glucose ≥180 mg/dL and HbA1c ≥ 7.0% at Screening.
* Known or suspected hypersensitivity to the trial product or related products.
* Participation in any other clinical studies within 30 days prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-11-11 (Actual); Primary Completion 2023-02-21 (Actual); Study Completion 2023-04-21 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 3, 7, 14, and 28 days after study medication
  Change in functional outcomes as measured by NIHSS from its baseline value
Barthel Index (BI) | 3, 7, 14, and 28 days after study medication
  Change in functional outcomes as measured by BI from its baseline value

SECONDARY OUTCOMES:
Thrombocyte Aggregation Test (TAT) | 3, 7, 14, and 28 days after study medication
  Change in haemostatic parameter as measured by TAT from its baseline value
Fibrinogen level | 3, 7, 14, and 28 days after study medication
  Change in haemostatic parameter as measured by fibrinogen level from its baseline value
D-dimer level | 3, 7, 14, and 28 days after study medication
  Change in haemostatic parameter as measured by d-dimer level from its baseline value
Liver function | 7 and 28 days after study medication
  Liver function measured includes: serum AST, ALT, gamma-GT, total bilirubin
Renal function | 7 and 28 days after study medication
  Renal function measured includes: serum creatinine
Routine hematology | 7 and 28 days after study medication
  Routine hematology measured includes: hemoglobin, hematocrit, RBC, WBC, differentiation of WBC, and platelet count
Adverse events | 1 - 28 days
  Adverse events, including bleeding events, will be observed and carefully evaluated along the course of the study

CONTACTS AND LOCATIONS:
Overall Officials: Paulus Sugianto, Sp.S(K), Dr, MD, Study Chair — Indonesia's Neurologists Organization (Perdossi); Muh. Hamdan, Sp.S(K), MD, Principal Investigator — Neurology Department Dr. Soetomo Hospital; Dodik Tugasworo, Sp.S(K), MD, Study Director — Neurology Department Dr. Kariadi General Hospital; Dian Cahyani, Sp.S, MD, Principal Investigator — Neurology Department Budhi Asih Hospital; Diah H Soeryaningtias, Sp.S, MD, Principal Investigator — Neurology Department Haji Surabaya Hospital; Gotot S PW, Sp.S, MD, Principal Investigator — Neurology Department Pasar Rebo Hospital; Sugeng Wijayanto, Sp.S, MD, Principal Investigator — Neurology Department Sidoarjo Regional General Hospital; Ika Y Margaretha, Sp.S, MD, Principal Investigator — Neurology Department Fatmawati Regional General Hospital; Wiwin Sundawiyani, Sp.S, MD, Principal Investigator — Islam Jakarta Hospital (RSIJ) Cempaka Putih; Rivan Danuaji, Sp.N(K), MD, Principal Investigator — Neurology Department Dr. Moewardi Hospital; Hanindia R. Prabaningtyas, Sp.S(K), MD, Principal Investigator — Neurology Department Universitas Sebelas Maret (UNS) Hospital
Locations (10):
- Indonesia (10):
  - Neurology Department, Dr. Kariadi General Hospital, Semarang, Central Java
  - Universitas Sebelas Maret (UNS) Hospital, Sukoharjo, Central Java
  - Dr. Moewardi Hospital, Surakarta, Central Java
  - Neurology Department Fatmawati Regional General Hospital, Jakarta, DKI Jakarta
  - Neurology Department, Budhi Asih Hospital, Jakarta, DKI Jakarta
  - Neurology Department, Pasar Rebo Hospital, Jakarta, DKI Jakarta
  - Neurology Department Islam Jakarta Hospital (RSIJ) Cempaka Putih, Jakarta Pusat, DKI Jakarta
  - Neurology Department Sidoarjo Regional General Hospital, Sidoarjo, East Java
  - Neurology Department, Haji Surabaya Hospital, Surabaya, East Java
  - Stroke/Cerebrobascular Division, Neurology Department, Dr. Soetomo Hospital, Surabaya, East Java